CLINICAL TRIAL: NCT02810184
Title: Determination of Bone Volume Changes of the Cranial Bone-augmented Jaw: A Feasibility Study
Acronym: VOLCRAN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Johan Abeloos, Head of department, Division of Maxillofacial surgery, AZ Sint-Jan AV
Other Study IDs: B049201627591
Record Dates: First submitted 2016-06-13; First posted 2016-06-22 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Severely Atrophic Jaw
Keywords: bone augmentation; long-term bone volume changes; immediate provisional implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CBCT arm: all participating patients receive an additional CBCT scan at 24 and 36 months, for analysis of evolution of bone volume
  Interventions: Radiation: cone-beam computed tomography (CBCT)

INTERVENTIONS:
Radiation: cone-beam computed tomography (CBCT) — additional CBCT scan at 24 and 36 months, for analysis of evolution of bone volume

SUMMARY:
The investigators aim to determine the level of total bone volume remodeling at 6, 24 and 36 months post-surgery in patients who underwent immediate prosthetic rehabilitation through a cranial bone-grafted maxilla in combination with immediate provisional implant (IPI) placement.

DETAILED DESCRIPTION:
Background

Bone augmentation provides a solution for patients with a severely atrophic jaw to achieve immediate fixed prosthetic rehabilitation. Studies reporting total bone volume changes are lacking.

Objectives

The investigators aim to determine the level of total bone volume remodeling at 6, 24 and 36 months post-surgery in patients who underwent immediate prosthetic rehabilitation through a cranial bone-grafted maxilla in combination with immediate provisional implant (IPI) placement.

Study design

A prospective, longitudinal study.

All patients will be recruited at time of pre-surgical consultation.

During the surgical procedure, autogenous cranial graft reconstruction of the jaw is carried out under general anaesthesia.

Cone-beam CT (CBCT) scans (NewTom VGi evo, QR Verona, Italy) will be taken pre-operatively, and at different time-points post-operatively to evaluate the remodeling process of the bone after the grafting procedure with implant placements and assess the total bone volume changes up to 3 years post-surgically.

CBCT scans will be send to the oral maxillofacial surgery (OMFS) Research Group within the Department of Imaging and Pathology (IMPATH), Catholic University Leuven (liaised with the clinical department of Oral and Maxillofacial Surgery; University Hospital Leuven) for analysis of the total bone volume.

Data related to patient demographics, clinical diagnosis, the surgical procedure, IPI stability, and total bone volume at different time-points will be registered by a clinical research coordinator.

Conclusion

This prospective trial could add important knowledge to the field, and provide indications to improve future clinical pre-prosthetic management.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages
* Patients with moderate to extreme bone atrophy of the jaw (class IV to VI according to Cawood and Howell (Cawood & Howell, 1988), caused by terminal periodontitis or edentulism
* Patients requiring bone augmentation procedures through cranial bone-grafting for jaw reconstruction
* Patients requesting immediate prosthetic rehabilitation, through the placement of an immediate provisional implant (IPI)-supported fixed bridge (immediate loading)

Exclusion Criteria:

* Patients not fulfilling abovementioned criteria
* Patients with severe uncontrollable diabetes
* Patients with a smoking habit of >10 cigarettes/day
* Patients with severe sinusitis problems
* Patients with insufficient cranial bone thickness
* Patients with bone remodeling or systemic diseases, or undergoing systematically administered treatments affecting bone remodeling
* Patients in whom postoperative complications (e.g. sinusitis, infections) occurred, will be excluded from the analysis, since these could be responsible for short-term bone volume loss confounding long-term results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06; Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
mean total bone volume changes (%) | 6, 24, and 36 months post surgery

SECONDARY OUTCOMES:
correlation between biologic risk factors, as collected through medical files and patient interview, with undesirable bone volume changes | short-term (6 months)
correlation between biologic risk factors, as collected through medical files and patient interview, with undesirable bone volume changes | long-term (24 months)
correlation between biologic risk factors, as collected through medical files and patient interview, with undesirable bone volume changes | long-term (36 months)
correlation between mechanical risk factors, as measured through clinical or radiographical visualization by the treating surgeon and/or prosthodontist, with undesirable bone volume changes | short-term (6 months)
correlation between mechanical risk factors, as measured through clinical or radiographical visualization by the treating surgeon and/or prosthodontist, with undesirable bone volume changes | long-term (24 months)
correlation between mechanical risk factors, as measured through clinical or radiographical visualization by the treating surgeon and/or prosthodontist, with undesirable bone volume changes | long-term (36 months)
incidence of immediate provisional implants loss | up to 6 months
incidence of definitive implant loss | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Johan Abeloos, MD, PhD, Principal Investigator — Head of Department
Locations (1):
- Division of Maxillofacial Surgery, Department of Surgery, AZ Sint-Jan Brugge-Oostende AV, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No